CLINICAL TRIAL: NCT02646501
Title: Prospective Randomized Clinical Trial for Effect of Stellate Ganglion Block in Medically Refractory Ventricular Tachycardia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0743
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Refractory Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A+PSGB (Experimental): (Antiarrhythmic drug + percutaneous stellate ganglion block) group
  Interventions: Drug: Antiarrhythmic drug; Procedure: percutaneous stellate ganglion block (PSGB)
- group A (Active Comparator): Antiarrhythmic drug group
  Interventions: Drug: Antiarrhythmic drug

INTERVENTIONS:
Drug: Antiarrhythmic drug — Antiarrhythmic drug
Procedure: percutaneous stellate ganglion block (PSGB) — percutaneous stellate ganglion block (PSGB)
  Arms: group A+PSGB

SUMMARY:
The investigators will compare the effects of PSGB(percutaneous stellate ganglion block) in patients with recurrent sustained VT/VF in spite of appropriate medical therapy and cardio-version/ defibrillation after correction of underlying correctable factors with those without PSGB by prospective randomized trail. PSGB will be performed every 3 days by anesthesiology specialist after cardiologist's request, until the stabilization of VT/VF. We will compare the frequency and episode number of VT/VF, procedure related complication, acute and long-term mortality.

DETAILED DESCRIPTION:
Recurrent ventricular tachycardia(VT)/ fibrillation(VF) increases mortality, especially in patients with structural heart disease. It has been reported that cardiac sympathectomy reduces VT/VF episodes in patients with complex VT, long QT syndrome, catecholaminergic polymorphic VT, or myocarditis. However, cardiac sympathectomy operation is hard to conduct in patients with hemodynamically unstable recurrent VT/VF or electrical storm. Therefore, we hypothesized that bed-side percutaneous stellate ganglion block (PSGB) reduces VT/VF episodes and mortality in patients with repetitive VT/VF who are properly managed with optimal medical therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients agreement of consent
* AF patient age 20-85
* Patient are diagnosed Refractory Ventricular tachycardia
* Patients who have generated Refractory Ventricular tachycardia despite of defibrillation and drug therapy
* Patients with ICD have generated ICD shock or anti-tachycardia pacing despite of defibrillation and drug therapy

Exclusion Criteria:

* Patients who do not agree with study inclusion
* Patients who do not taken stellate ganglion block due to unstable hemodynamic status
* Patients have experienced major hemorrhagic complication
* Patients of the DNR status
* Patients with malignancy tumor, major neurogenic disease or gastrointestinal disease

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Number of VT/VF episodes after randomization | 5 days after randomization
Duration of VT/VF episodes after randomization | 5 days after randomization

SECONDARY OUTCOMES:
mortality | 1 month after the enrollment
  death, cause of death,
procedure related complication | 1 month after the enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No